CLINICAL TRIAL: NCT02007005
Title: Dose-Escalation-Study With abnobaVISCUM® Fraxini 2 (AVF2) as Intravesical Instillation in Patients With Superficial Bladder Cancer According to ICH/GCP (International Conference on Harmonisation/Good Clinical Practice) - Guidelines: a Phase Ib/IIa Study
Brief Title: Maximum Tolerable Concentration of abnobaVISCUM Fraxini Intravesically in Patients With Superficial Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abnoba Gmbh (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB01
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Superficial Bladder Cancer
Keywords: superficial bladder cancer; mistletoe extract; maximum tolerated dose; marker tumor; remission; recurrence rate
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — viscum album peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalation (Experimental): intravesical instillation of abnobaVISCUM Fraxini
  Interventions: Drug: abnobaVISCUM Fraxini

INTERVENTIONS:
Drug: abnobaVISCUM Fraxini — intravesical instillation 6 times, once weekly, in increasing dosages until dose-limiting-toxicity occurs
  Other Names: viscum album extract; mistletoe extract; abnobaVISCUM

SUMMARY:
The aim of this phase Ib/IIa study is to investigate the maximum tolerable concentration of abnobaVISCUM® Fraxini for intravesical instillation in patients with superficial bladder cancer. Secondary objectives are the local and systemic tolerability, the influence on tumor remission and the influence on the one-year recurrence rate.

DETAILED DESCRIPTION:
A dose-escalation-study according ICH/GCP (International Conference on Harmonisation/Good Clinical Practice) with different concentrations of abnobaVISCUM® Fraxini is conducted in two hospitals in Germany and Egypt. Patients with superficial bladder cancer TaG1/G2 or T1G1/G2 are enclosed after TUR-B (transurethral resection bladder). The tolerability of the different concentrations is assessed after weekly instillations into the urinary bladder for 6 weeks. A direct antitumoral effect is assessed on a single marker tumor left in the bladder after a complete TUR of all other lesions according a study design established by the EORTC-GENITO-URINARY GROUP (European Organisation for Research and Treatment of Cancer). A re-TUR is conducted after 12 weeks. Tumor response is measured by biopsy of the marker lesion and by cytology. Safety of the instillations is measured by analysis of adverse events, vital signs and clinical laboratory tests. After treatment of a cohort is finished a safety evaluation is conducted to decide about the increase to the next dosage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically proved superficial bladder cancer (Ta G1/G2 or T1G1/G2) 2 - 7 weeks before transurethral resection
* Written informed consent for study participation and for documentation of disease data including further distribution of these data

Exclusion Criteria:

* Muscle invasive bladder carcinoma and/or carcinoma in situ (CIS)
* Intravesical instillation therapy within 6 months prior to study enrolment
* Radiotherapy of the bladder prior to study enrolment
* Contracted bladder (capacity less than 100 ml)
* Non treated acute or chronic urinary tract infection
* Allergy against mistletoe extract preparations
* Subvesical obstructions (e. g. prostate hyperplasia, urethral stenosis, residual urine volume more than 80 ml)
* Severe illnesses and circumstances not permitting study participation (e. g. alcoholism or substance abuse)
* Pregnancy or lactation (pregnancy test if required) as well as women without sufficient contraception
* Participation in another clinical study within 30 days prior to this study
* Administration of immunotherapeutic and/or cytostatic drugs within 4 weeks prior to study enrolment
* Chronic progressive infections (e. g. tuberculosis)
* Pre-treatment with mistletoe extracts/mistletoe lectins

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-01; Primary Completion 2012-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerable concentration of abnobaVISCUM Fraxini for intravesical instillation | 6 weeks
  The primary objective is to investigate the maximum tolerable concentration of abnobaVISCUM Fraxini for intravesical instillation in patients with superficial bladder cancer. The treatment schedule included 6 weekly instillations.

SECONDARY OUTCOMES:
Local and systemic tolerability of different concentrations of abnobaVISCUM Fraxini for intravesical instillation | 6 weeks
  Secondary objectives are to investigate the local and systemic tolerability of different concentrations of abnobaVISCUM Fraxini for intravesical instillation. Main variables of safety analysis are adverse events, vital signs and clinical laboratory tests.
Influence on remission and influence on the one year recurrence rate of abnobaVISCUM Fraxini for intravesical instillation | up to 1 year
  Secondary objectives are to investigate the influence on remission and influence on the one year recurrence rate measured by histological examination of biopsies of the marker lesion, cytology and cystoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Ruebben, Prof.Dr.Dr., Study Director — Director of the Urological Clinic of the University Hospital Essen
Locations (2):
- Theodor Bilharz Research Institute, Giza, Egypt
- Clinic of Urology of the University Hospital of Essen, Essen, Germany

REFERENCES:
- [Result] Rose A, El-Leithy T, vom Dorp F, Zakaria A, Eisenhardt A, Tschirdewahn S, Rubben H. Mistletoe Plant Extract in Patients with Nonmuscle Invasive Bladder Cancer: Results of a Phase Ib/IIa Single Group Dose Escalation Study. J Urol. 2015 Oct;194(4):939-43. doi: 10.1016/j.juro.2015.04.073. Epub 2015 Apr 22. PMID 25910967